CLINICAL TRIAL: NCT02161237
Title: A Multi-center, Randomized, Open-label, Pilot and Exploratory Study Investigating Safety and Efficacy in OPTIMIZEd Dosing of Advagraf® Kidney Transplantation in Asia.
Brief Title: Asian Study to Investigate Safety and Efficacy of Optimized Dosing of Advagraf in Kidney Transplantation
Acronym: OPTIMIZE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 506-MA-1001
Record Dates: First submitted 2014-06-09; First posted 2014-06-11 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Kidney Transplantation
Keywords: Acute rejection; Advagraf; Renal function
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard dose group (Experimental): Oral
  Interventions: Drug: Advagraf®
- optimized dose group (Experimental): Oral
  Interventions: Drug: Advagraf®

INTERVENTIONS:
Drug: Advagraf® — oral
  Other Names: FK506; tacrolimus

SUMMARY:
Primary purpose of this study is to compare renal function between subjects receiving optimized dose Advagraf® over 52 weeks after kidney transplantation and subjects receiving standard dose Advagraf®. Pilot results of safety and efficacy in optimized dose Advagraf® over 52 weeks after kidney transplantation will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* End stage kidney disease and a suitable candidate for primary kidney transplantation or re-transplantation
* Receiving a kidney transplant from a deceased or living donor with compatible ABO blood type
* Female subject of childbearing potential must have a negative serum pregnancy test at enrollment and must agree to maintain effective birth control during the study. And, male subject of childbearing potential should agree to maintain effective birth control during the study

Exclusion Criteria:

* Receiving or having previously received an organ transplant other than a kidney
* Cold ischemia time of the donor kidney > 24 hours
* Receiving a graft from a non-heart-beating donor other than of Maastricht category 3
* Significant liver disease
* Receiving a graft from a hepatitis C or B positive donor
* Requiring on-going dosing with a systemic immunosuppressive drug prior to transplantation (e.g. for Lupus disease, FSGN etc) other than minimal levels of immunosuppressant following failure of a previous transplantation without nephrectomy
* Significant, uncontrolled concomitant infections and/or severe diarrhea, vomiting, active upper gastro-intestinal tract mal absorption or active peptic ulcer
* Subject or donor known to be HIV positive
* Known allergy or intolerance to tacrolimus, macrolide antibiotics, steroids, lactose, basiliximab or MMF or any of the product excipient
* Subject has malignant tumor
* Currently participating in another clinical trial, and/or has taken an investigational drug within 12 weeks prior to the study
* Subject with a high immunological risk

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2014-06-26 (Actual); Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
estimated GFR | at Week-52 after transplantation

SECONDARY OUTCOMES:
creatinine clearance | at Week-52 after transplantation
serum creatinine level | at Week-52 after transplantation
Number of graft survival | at Week-52 after transplantation
Subject survival | at Week-52 after transplantation
number of biopsy-proven acute rejection | at Week-52 after transplantation
Composite of graft loss, subject death and biopsy proven acute rejection | at Week-52 after transplantation
Time to the first acute rejection | up to Week-52 after transplantation
Time to the first steroid-resistant acute rejection | up to Week-52 after transplantation
Severity of biopsy proven acute rejection | up to Week-52 after transplantation
  Severity is evaluated using Banff '07 Criteria
Safety assessed by the incidence of adverse events, vital signs and lab tests | for 52 weeks after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (2):
- Seoul, South Korea
- Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=233